CLINICAL TRIAL: NCT01742780
Title: A Study Evaluating Insertion Site Identification Methods Used to Establish Intraosseous Vascular Access in the Proximal Humerus
Brief Title: Evaluation of Various Methods Used to Identify the Proximal Humerus Intraosseous Vascular Access Site
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2012-16
Record Dates: First submitted 2012-11-30; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Proximal Humerus Intraosseous Vascular Access
Keywords: Intraosseous Vascular Access; IO Access; IO Vascular Access; EZ-IO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard Vidacare Site Identification Method (Active Comparator): Palpate up the proximal humerus towards the anterior shoulder just above the surgical neck, to the greater tubercle of the proximal humerus. Insert the needle set perpendicular to skin with a slight downward angle at the most prominent aspect of greater tubercle to establish proximal humerus intraosseous vascular access.
  Interventions: Procedure: Proximal Humerus Intraosseous Vascular Access
- Saussy Site Identification Method (Active Comparator): Palpate the proximal humerus to locate the intertubercular groove; rotate the forearm medially and laterally to isolate the groove. Move one finger breadth laterally from the groove to the greater tubercle. Insert perpendicular to skin with a slight downward angle to establish proximal humerus intraosseous vascular access.
  Interventions: Procedure: Proximal Humerus Intraosseous Vascular Access
- Campbell Site Identification Method (Active Comparator): With the fingers on both hands fully extended similar to a karate chop, place one hand into the anterior joint space (acromioclavicular joint) of the patient. Place the second "karate chop" hand along the midline of the patient's lateral shoulder; touch the pinkie fingers over the superior aspect of the patient's shoulder. Overlap the thumbs on the patient's shoulder, which will be at the most prominent aspect of the greater tubercle. Insert the needle set perpendicular to skin with a slight downward angle to establish proximal humerus intraosseous vascular access.
  Interventions: Procedure: Proximal Humerus Intraosseous Vascular Access
- Davlantes Site Identification Method (Active Comparator): Using one hand, place the thumb on the acromioclavicular joint in the natural recess or "pocket" between the distal clavicle and the humeral head, wrapping the rest of the hand around the upper arm. The hand should be oriented such that the index finger and rest of the hand is at a 90-degree angle to the thumb. The webspace between the thumb and index finger will be approximately where the surgical neck of the humerus is; move one finger breadth (approximately 1 cm) superior. Insert perpendicular to skin with a slight downward angle to establish proximal humerus intraosseous vascular access.
  Interventions: Procedure: Proximal Humerus Intraosseous Vascular Access

INTERVENTIONS:
Procedure: Proximal Humerus Intraosseous Vascular Access — EZ-IO Intraosseous Vascular Access System
  Other Names: EZ-IO proximal humerus intraosseous vascular access

SUMMARY:
The purpose of this study is to determine if there is one method of identifying the proximal humerus intraosseous vascular access site that is easier for clinicians to use, out of the 4 methods being evaluated.

ELIGIBILITY:
Inclusion Criteria Device Operators:

* Recent/current experience in the medical field as a practicing clinician.
* Currently licensed/certified Emergency Medicine Technician, paramedic, or nurse
* Have had no formal training on use of the proximal humerus intraosseous insertion site.

Exclusion Criteria Device Operators:

There is no exclusion criteria

Inclusion Criteria Healthy Volunteers

* Age 21 years or older.
* Has no amputation of the upper extremities.
* Able to lay flat on table for up to 2 hours.
* Self-reported as healthy.

Exclusion Criteria Healthy Volunteers:

* Have an active infection in the body
* Imprisoned
* Pregnant
* Cognitively impaired
* Fracture in humerus, or significant trauma to the site
* Excessive tissue and/or absence of adequate anatomical landmarks in humerus
* Infection in target area
* Humeral intraosseous insertion in past 48 hours, prosthetic limb or joint or other significant orthopedic procedure in humerus
* Current use of anti-coagulants

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Ease of use score | Within 10 minutes of procedure
  Device operators will complete an ease of use questionnaire regarding the assigned site identification method.
Level of confidence score | within 10 minutes of procedure
  Device operators will complete a level of confidence questionnaire regarding their assigned site identification method.
Site identification success/failure | within 10 minutes of the procedure
  The ability of the device operator to identify the proximal humerus intraosseous insertion site will be graded as success or failure.
Time to intraosseous catheter placement | within 10 minutes of the procedure
  The amount of time it takes for the device operator to identify the proximal humerus intraosseous insertion site and insert the needle.

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Miller, MD, Principal Investigator — Vidacare Corporation
Locations (1):
- Bulverde-Spring Branch EMS, Spring Branch, Texas, United States

REFERENCES:
- [Background] Reades R, Studnek JR, Vandeventer S, Garrett J. Intraosseous versus intravenous vascular access during out-of-hospital cardiac arrest: a randomized controlled trial. Ann Emerg Med. 2011 Dec;58(6):509-16. doi: 10.1016/j.annemergmed.2011.07.020. PMID 21856044
- [Background] Reades R, Studnek JR, Garrett JS, Vandeventer S, Blackwell T. Comparison of first-attempt success between tibial and humeral intraosseous insertions during out-of-hospital cardiac arrest. Prehosp Emerg Care. 2011 Apr-Jun;15(2):278-81. doi: 10.3109/10903127.2010.545479. Epub 2011 Jan 28. PMID 21275573
- [Background] Wampler D, Schwartz D, Shumaker J, Bolleter S, Beckett R, Manifold C. Paramedics successfully perform humeral EZ-IO intraosseous access in adult out-of-hospital cardiac arrest patients. Am J Emerg Med. 2012 Sep;30(7):1095-9. doi: 10.1016/j.ajem.2011.07.010. Epub 2011 Oct 24. PMID 22030185